CLINICAL TRIAL: NCT05771363
Title: Frequency and Risk Factors for Autoimmune Disorders and Rheumatic Manifestations in Egyptian Patients With Inflammatory Bowel Disease
Brief Title: Frequency and Risk Factors for Autoimmune Disorders and Rheumatic Manifestations in Egyptian Patients With IBD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amaal fathi mousa ali, physician, Assiut University
Other Study IDs: rheumatology in IBD
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: IBD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To examine the prevelance of autoimmune disorders and rheumatic manifestations in egyptian patients with inflammatory bowel diseases,and asses the relation between prevelance of autoimmune disorders ,rheumatic manifestations and disease activity of IBD

ELIGIBILITY:
Inclusion Criteria:

* 1-adult patients with adiagnosis of IBD according to the validated criteria. 2-patients>18 years without aprevious diagnosis of SPA or other rheumatological manifestations.

Exclusion Criteria:

* 1- patients with active cancer or lymphoproliferative disease. 2-patients with uncontrolled diabetes. 3-patients with unstable ischeamic heart disease or congestive heart failure. 4-patients with acute renal failure. 5-patients already diagnosed with inflammatory or crystal induced arthropathies (including gout and calcium pyrophosphate dehydrate deposition disease) or other autoimmune diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cross-sectional studies are observational studies that analyze data from a population at a single point in time. They are often used to measure the prevalence of health outcomes, understand determinants of health, and describe features of a population. Unlike other types of observational studies, cross-sectional studies do not follow individuals up over time. They are usually inexpensive and easy to conduct. They are useful for establishing preliminary evidence in planning a future advanced study. This article reviews the essential characteristics, describes strengths and weaknesses, discusses methodological issues, and gives our recommendations on design and statistical analysis for cross-sectional studies in pulmonary and critical care medicine. A list of considerations for reviewers is also provided.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
frequency and risk factors for autoimmune disorders and rheumatic manifestations in Egyptian patients with inflammatory bowel diseases. | 1year
  to examine the prevelance of autoimmune disorders and rheumatological manifestations in Egyptian patients with inflammatory bowel diseases

REFERENCES:
- [Background] Lanna CC, Ferrari Mde L, Rocha SL, Nascimento E, de Carvalho MA, da Cunha AS. A cross-sectional study of 130 Brazilian patients with Crohn's disease and ulcerative colitis: analysis of articular and ophthalmologic manifestations. Clin Rheumatol. 2008 Apr;27(4):503-9. doi: 10.1007/s10067-007-0797-5. Epub 2007 Dec 21. PMID 18097711